CLINICAL TRIAL: NCT01141504
Title: Effect of Oral ATP on Human Muscle Performance
Brief Title: Effect of Oral Adenosine-triphosphate (ATP) on Human Muscle Performance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Metabolic Technologies Inc. (Industry)
Collaborators: Iowa State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: MTI2010-CS01
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Healthy Subjects
Keywords: Supplemental ATP; Muscle Work Performed; Muscle Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Oral placebo capsules similar in color and size to the intervention
  Interventions: Dietary Supplement: Placebo
- PeakATP 250 (Active Comparator): Oral supplement capsules containing 250 mg/day of PeakATP
  Interventions: Dietary Supplement: PeakATP 250
- PeakATP 400 (Active Comparator): Oral supplement capsules containing 400 mg/day of PeakATP
  Interventions: Dietary Supplement: PeakATP 400
- PeakATP 400 plus proprietary blend (Active Comparator): Oral supplement capsules containing 400 mg/day of PeakATP plus a proprietary blend
  Interventions: Dietary Supplement: PeakATP 400 plus proprietary blend

INTERVENTIONS:
Dietary Supplement: PeakATP 250 — The nutritional intervention provides for oral ingestion of 250 mg PeakATP per day
  Arms: PeakATP 250
Dietary Supplement: Placebo — Placebo capsules that are comparable in size and color to the active comparator for blinding purposes
  Arms: Placebo
Dietary Supplement: PeakATP 400 — The nutritional intervention provides for oral ingestion of 400 mg PeakATP per day
  Arms: PeakATP 400
Dietary Supplement: PeakATP 400 plus proprietary blend — The nutritional intervention provides for oral ingestion of 400 mg PeakATP per day plus a proprietary blend of additional nutrients
  Arms: PeakATP 400 plus proprietary blend

SUMMARY:
Adenosine-triphosphate (ATP) serves as the sole energy source for muscle contraction. Therefore human performance of brief maximal exercise is limited, in part, by the availability of ATP to the contracting muscle. Because muscle ATP storage is small (enough to sustain maximal exercise for less than 1 second), factors that enhance either storage or resynthesis of ATP may have a positive impact on repeated muscle contractions. The current study will test the hypothesis that increasing ATP availability to muscle via oral supplementation will improve performance of repeated high intensity exercise as measured by a) work performed in each of the three 50 contraction fatigue tests, b) sum of total work performed, and c) percentage decrement in total work from the first to third third 50 contraction test.

DETAILED DESCRIPTION:
To date we have studied 10 subjects who have followed through with all 3 of the original interventions (Placebo, 250 mg PeakATP/d and 400 mg PeakATP/d). Currently we have received approval and are expanding the study with 5 additional subjects who will receive the Placebo, 400 mg PeakATP/d and the 400 mg PealATP/d plus proprietary blend interventions.

ELIGIBILITY:
Inclusion Criteria:

* No major medical conditions;
* Able to perform fatigue testing procedures;
* Not currently taking prescription medications;
* Not currently taking dietary supplements (a daily multi-vitamin not exceeding RDA is permitted)

Exclusion Criteria:

* Major medical condition affecting metabolism or general function;
* Not able to perform fatigue testing;
* Taking prescription medications;
* Taking a dietary supplement other than a multi-vitamin not exceeding RDA

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Work Performed | Measured after 15 days of intervention
  The work and total work performed in 3 exercise fatigue tests given after 15 days of nutritional intervention.

SECONDARY OUTCOMES:
Decrease in work performed in each successive test | Measured after 15 days of intervention
  The decrease in total work performed in each of 3 successive fatigue tests will be measured and used as a measure of muscle fatigability after 15 days of nutritional intervention

CONTACTS AND LOCATIONS:
Overall Officials: John A Rathmacher, PhD, Principal Investigator — Metabolic Technologies Inc.
Locations (1):
- Iowa State University, Ames, Iowa, United States